CLINICAL TRIAL: NCT02594917
Title: Genetic and Environmental Determinants That Control Metabolism in Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Stephen Y. Chan, Associate Professor of Medicine, University of Pittsburgh
Other Study IDs: STUDY19030124
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Iron-sulfur Cluster Deficiency; Pulmonary Hypertension; Friedreich Ataxia
MeSH Terms: conditions — Hypertension, Pulmonary; Friedreich Ataxia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are generating inducible pluripotent stem cells from blood and skin biopsies from participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test Group: The study population will include ten patients (ages 18-60 yrs) with confirmed mutations of the iron-sulfur cluster biogenesis complex of proteins and experiencing dyspnea, heart failure, or exercise intolerance.
  Interventions: Procedure: Right Heart Catheterization; Other: Blood draw
- Control Group: It will also include ten additional patients (ages 18-60 yrs) who are unaffected first-degree family members of the above subjects.
  Interventions: Other: Blood draw

INTERVENTIONS:
Procedure: Right Heart Catheterization — Some participants (i.e., those that are willing and able) will undergo a Right Heart Catheterization to check Cardiopulmonary function.
  Groups: Test Group
Other: Blood draw — Test and control group will be asked to give 20 ml of blood samples

SUMMARY:
The investigators are performing this research study to determine whether having low iron-sulfur cluster levels can cause a disease known as pulmonary hypertension (PH). PH is defined as abnormally high blood pressure in the arteries of the lungs.

Usually, small specialized structures inside each human cell called mitochondria are in charge of generating energy within lung arteries for normal function. During situations of disease or stress, lung arteries undergo a change in the function of mitochondria, resulting in the development of PH. In studies on mice, investigators have learned that alterations in the production of specific metal complexes called iron-sulfur clusters are responsible for these changes. This makes it more likely that mice will develop PH.

In this study, the investigators want to find out if alteration of iron-sulfur cluster formation leads to increased likelihood of developing PH in humans.

DETAILED DESCRIPTION:
Test group:

The study will include two visits for the test group:

At visit one there will be required and optional research activities as the following:

Required research activities:

-Peripheral blood draw (3.5 tablespoons) drawn by research coordinator. This blood is to isolate PBMCs for generation of iPSCs.If patient did not want to give a blood sample we will ask if willing to give a urine sample. A clinical research coordinator will give the patient a plastic container and will explain how use it.

The following research activities will be optional at visit one:

1. Physical exam and blood work (kidney/liver, blood count, coagulation, B-HCG, iron studies, and plasma for microRNA) processed at Presby Lab. This will be required if the patient approved to do right heart cath.
2. Electrocardiogram.
3. 6 Minute Walk Test.
4. Skin Biopsy from underarm or inner thigh by physician (Dermatology department) (if patients agree to do, if not, we will only get a blood sample)
5. Resting Echocardiogram

This visit will last 7-8 hours.

Study Visit Two:

This will include optional Right Heart Catheterization.

* Right Heart catheterization by PI/Sub-Investigator. Duration ~ 3 hours

  * IF the results show that the pressure in the lung vessels is elevated without exercise AND there is no other abnormality in the heart function, we will NOT do exercise testing.
  * IF the patients are physically able to perform exercise testing/agree to do an exercise testing, patients will have an Exercise Right Heart catheterization and a Rest and Stress Echocardiography. (Determined by PI/Sub-Investigator
  * All participants who will do right heart catheterization will have to do a pregnancy test before the procedure.
* Exercise Echocardiogram completed in. If patient unable to exercise medication (Dobutamine) will be given. Duration ~ 1-2 hours
* Exercise Right Heart catheterization Duration ~ 2-3 hours

CONTROL GROUP

Control group will only have one visit. At this visit there will be a minimum required research activity to participate in the study and this will include:

-Peripheral blood draw (3.5 tablespoons) drawn by research coordinator. This blood is to isolate PBMCs for generation of iPSCs. If participant did not want to give a blood sample we will ask if willing to give a urine sample.

The following research activists will be optional at visit one:

1. Physical exam and blood work (kidney/liver, blood count, coagulation, B-HCG, iron studies, and plasma for microRNA) processed at Presby Lab. This will be required if the patient approved to do right heart cath.
2. ECG, done by research coordinator and read by PI/Sub-Investigator.
3. 6 Minute Walk Test, done by research coordinator, if patient could perform.
4. Skin Biopsy from underarm or inner thigh by physician (Dermatology department) (if patients agree to do, if not, we will only get a blood sample) This visit will last 6-7 hours.

ELIGIBILITY:
INCLUSION CRITERIA for Test Group:

1. Consenting individuals age 18-60 years of age
2. Have a confirmed genetic homozygous mutation (including ISCU1/2, FXN, BOLA3, NFU1) that causes the impairment of iron-sulfur cluster formation; such a subject will not be excluded from this study even if that patient's first degree relative(s) does not enroll in this pilot study.

INCLUSION CRITERIA for Control Group:

1. Consenting individuals age 18-60 years of age
2. First degree family member (mother, father, sister, brother, son, or daughter) of recruited individual in the test group
3. Have a confirmed heterozygous genetic mutation (including ISCU1/2, FXN, BOLA3, NFU1)

EXCLUSION CRITERIA for Test and Control Group:

1. Impaired decision making capacity
2. Inability to consent to procedures
3. Children less than 18 years of age and adults older than 60 years of age
4. Current pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will include ten patients (ages 18-60 yrs) with confirmed mutations of the iron-sulfur cluster biogenesis complex of proteins. It will also include ten additional patients (ages 18-60 yrs) who are unaffected first-degree family members of the above subjects.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
6 minute walk distance (meters) | baseline
  In the TEST group, the investigators will measure 6 minute walk distance
Pulmonary arterial pressure (mm Hg) | baseline
  In the TEST group, the investigators will measure pulmonary arterial pressure by right heart catheterization at rest and with exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chan, MD, PhD, FAHA, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided